CLINICAL TRIAL: NCT03308253
Title: Pilot Study for Antibiotic Impregnated Calcium Sulfate Beads as Prophylaxis for Surgical Site Infection in Vascular Surgery Patients
Brief Title: Study for Antibiotic Impregnated Calcium Sulfate Beads as Prophylaxis for Surgical Site Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Antimicrobial Beads
Record Dates: First submitted 2017-10-03; First posted 2017-10-12 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Surgical Site Infection
Keywords: Vascular Surgery; Surgical Site Infection; Prophylactic Antibiotics; Implantable Beads
MeSH Terms: conditions — Surgical Wound Infection | interventions — Vancomycin; Tobramycin; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Other): Patients will receive the standard of care for vascular procedures as it is provided at Hamilton General Hospital
  Interventions: Other: Standard of Care
- Antibiotic Impregnated Beads (Experimental): Patients will have their wound packed with calcium sulfate beads prior to closing. The beads will be infused with the antibiotics vancomycin and tobramycin.
  Interventions: Device: Stimulan Rapid Cure; Drug: Vancomycin; Drug: Tobramycin

INTERVENTIONS:
Device: Stimulan Rapid Cure — Calcium sulfate dissolvable beads
  Arms: Antibiotic Impregnated Beads
Drug: Vancomycin — 0.5 g Vancomycin per patient
  Arms: Antibiotic Impregnated Beads
Drug: Tobramycin — 120 mg tobramycin per patient
  Arms: Antibiotic Impregnated Beads
Other: Standard of Care — Standard of care provided at Hamilton General Hospital consisting of dressings for the wound.
  Arms: Standard of Care

SUMMARY:
The CDC quotes a rate of wound infection of 2-5% for inpatient surgery. Patients undergoing a vascular operation, however, are generally at an increased risk of wound infection with rates often close to 5-10%. Groin incisions are an additional risk factor for surgical site infections, with rates of wound infection being quoted from 10-15%, and even as high as 30% in high risk patients. The use of implantable calcium sulfate beads mixed with antibiotics may help to lower the rate of infection in these high risk patients.

DETAILED DESCRIPTION:
The initial pilot will consist of 30 patients per arm and will provide estimates of effect size, event rates, and recruitment rates. It will mirror the final study in terms of methodology. This will occur at the Hamilton General Hospital (Hamilton, ON. Canada)

Patients will be randomized to either the exposure group or control group by the study coordinator. Patients will be block randomized among surgeons (6), so that each surgeon has an equal number of patients in the control and exposure arms. Randomization will occur once an operative date has been booked for a patient. The arm they are assigned to will be how the patient is treated, regardless of if they are cancelled and re-booked. Should patients be done as an emergency procedure, prior to their index procedure (when the beads would be implanted), they will be excluded from the study. As no intervention has occurred at this point, there will be no informative loss to follow-up or censoring and therefore this will not impact validity of the design. We are unable to provide beads for emergency procedures, as the research pharmacy is not open.

The research coordinator will inform the research pharmacy to produce calcium sulfate beads impregnated with Vancomycin (1g) and Tobramycin (240mg) for the exposure arm. The control arm will receive standard care. The only difference between standard care and the treatment arm is the use of the antibiotic calcium sulfate beads. Beads will be delivered in a sterile manner to the OR. For each patient half of a standard 10cc kit will be delivered (5cc of Stimulan Calcium Sulfate). As the beads are being applied only to a groin incision(s) this will provide an adequate volume of beads. It will also prevent insertion of excess beads.

Surgeons will insert the beads loosely within the soft tissue of groin incisions, so as not to distort the normal anatomy. This technique will be discussed with all surgeons prior to pilot initiation as a group. This will aim to standardize the method among involved surgeons. At the end of the study we will complete a focus group with surgeons to discuss their experience using the beads to better inform the protocol for the final RCT. Patients are randomized as a unit and therefore, if there are bilateral groin incisions, both will be treated as per their randomization.

Patients will be blinded to which treatment they receive. The beads are believed to be non-detectable to the patient. Only by means of wound dehiscence would a patient be expected to determine their treatment group. For practical reasons the surgeon cannot be blinded to treatment. Nurse assessors and study authors conducting review of patient records will be blinded to patient treatment.

Patients will be recruited from all patients consented for an included procedure at HGH. A study coordinator or a resident will obtain consent. The patient's primary physician will not be involved in the consent process.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged > 18
* Undergoing a revascularization procedure involving the femoral artery and requiring either unilateral or bilateral groin incision
* BMI > 30
* Presence of one of the following: current smoker, diabetes requiring pharmacologic intervention, previous re-vascularization procedure

Exclusion Criteria:

* Any patient with a current infection or requiring ongoing use of antibiotics
* Any patient who otherwise has an indication requiring the use of antibiotic impregnated material
* Known allergy or sensitivity to tobramycin or vancomycin
* Grade 4 or 5 chronic kidney disease
* Moderate or severe hypercalcemia
* Any woman currently pregnant or planning on becoming pregnant during the course of the study
* Any patient involved in another study that, in the investigators opinion, is believed will interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 30 days
  The primary outcome will be combined, superficial, deep or organ/space infection as defined by the CDC. The CDC definition for surgical site infection is one of the most widely used and is both the NSQUIP and NHSN definition.

SECONDARY OUTCOMES:
Wound Complication Rate | 30 day
  Wound complications will be defined as: wound dehiscence, skin edge necrosis, hematoma, seroma, increased wound exudate, graft exposure. These will be measured with a standardized form, by the blinded nurse assessor, at each follow-up appointment. They will additionally be assessed by the author reviewing patient records at thirty days. If imaging is required for diagnosis of hematoma or seroma, the result will be collected from the imaging records, and treated as consistent with the conclusions of the formal imaging report.
Surgical Graft Infection Rate | 90 day
  Graft infection is defined as; diagnosis by surgeon or surgical designate requiring re-operation or prolonged course of antibiotic therapy. An author blinded to patient treatment will review the records of the patient including patient charts, antibiotic prescriptions, home care and ID referrals and record the information in a standardized form for this endpoint.
Bacterial Resistance | 30 day
  In the event of infection requiring laboratory samples, screening for resistant bacteria will be performed. Bacterial cultures will be performed in order to determine the presence of tobramycin or vancomycin resistant strains.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Stacey, DS, Principal Investigator — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared for this pilot study.

REFERENCES:
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- [Derived] Cristino MA, Nakano LC, Vasconcelos V, Correia RM, Flumignan RL. Prevention of infection in aortic or aortoiliac peripheral arterial reconstruction. Cochrane Database Syst Rev. 2025 Apr 22;4(4):CD015192. doi: 10.1002/14651858.CD015192.pub2. PMID 40260835